CLINICAL TRIAL: NCT03692806
Title: A 3-month Randomized Double Blind Placebo-controlled Multicenter Study to Assess the Efficacy of STABLOR® on Visceral Fat Mass Reduction in Patients With Metabolic Syndrome
Brief Title: Efficacy of STABLOR® on Visceral Fat Mass Reduction in Patients With Metabolic Syndrome
Acronym: OBEMINALE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LNC THERAPEUTICS (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other); StatistiCal BV Wassenarr, The Netherland represented by Dr W.Calame (Unknown)
Responsible Party: Sponsor
Organization: YSOPIA Bioscience (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-A01402-53
Record Dates: First submitted 2018-09-10; First posted 2018-10-02 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stablor (Experimental): 2 sachets to be taken twice a day at breakfast and in the afternoon as a snack during 12 weeks
  Interventions: Dietary Supplement: Stablor
- placebo (Placebo Comparator): 2 sachets to be taken twice a day at breakfast and in the afternoon as a snack during 12 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Stablor — Stablor sachet
  Arms: Stablor
Dietary Supplement: placebo — placebo sachet
  Arms: placebo

SUMMARY:
The primary objective of the study is to assess the efficacy of STABLOR® consumption on visceral fat mass compared to placebo, in persons with metabolic syndrome during 12 weeks of consumption.

DETAILED DESCRIPTION:
It is expected that the food product STABLOR will reduce visceral fat mass in subjects with metabolic syndrome and therefore will improve cardiometabolic risk factors. The aim of the current study is to assess the impact of a 12-week intake of STABLOR, compared to a placebo, on visceral fat in patients with metabolic syndrome. The primary objective of the study is to assess the efficacy of 12-week STABLOR® consumption on visceral fat mass compared to placebo, in persons with metabolic syndrome. The Secondary outcomes include Anthropometric measurements and body composition, metabolic syndrome status, STABLOR® metabolism, Cardiovascular biomarkers, Systemic inflammation, Quality of life and Behavior.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* Age between 18 and 65 years (limits included),
* BMI between 27 and 40 kg/m² (limits included),
* With metabolic syndrome: Waist circumference > 94 cm for male (>90 cm for male of South-East Asian, Chinese and Japanese ethnic groups) and > 80 cm for female and at least two of the following criteria :

  * Triglycerides levels ≥ 1.5 g/L (1.71 mmol/L) or stable under treatment for at least 6 months,
  * HDL cholesterol levels <0.40 g/L (1.03 mmol/L) for male and <0.5 g/l (1.29 mmol/L) for female or stable under treatment for at least 6 months,
  * Fasting plasma glucose ≥1 g/L (5.6 mmol/L) and non-diabetic,
  * Blood pressure ≥130 mmHg (systolic) and/or 85 mmHg (diastolic) or stable under antihypertensive treatment for at least 6 months,
* Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,

Exclusion Criteria:

* Suffering from a metabolic disorder such as diabetes uncontrolled thyroidal trouble or other metabolic disorder,
* Suffering from a cardiac insufficiency, inflammatory disease, severe hepatic of renal insufficiency, or gastrointestinal disorders (Crohn's disease or Ulcerative Colitis) or others diseases found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease),
* Having suffered of stroke or ictus within the last 6 months,
* Suffering of depression,
* Had a major surgical procedure within the last 6 months,
* Had a bariatric surgery,
* With a known or suspected food allergy or intolerance to lactose or soja, or hypersensitivity to any of the study products' ingredient,
* Who does not like the investigational product flavors "vanilla-toffee", "chocolate" and "coffee",
* Having a biological selection profile considered as abnormal by the investigator (BUN, Creatinine, calcium, Liver enzymes (GGT, AST, ALT), Blood Cell Count, , HIV, HCV, lipids (TG, HDL, LDL, total cholesterol),glycaemia, B HCG),
* Pregnant (positive pregnancy test at selection visit) or lactating women or intending to become pregnant within 6 months ahead,
* Women of child bearing potential without efficient contraception,
* Under nutritional supplement or drugs acting on weight or satiety according to the investigator or stopped less than 6 months before the study,
* With a current or planned in the next 6 months specific diet (hypocaloric, vegan, vegetarian…) or stopped less than 6 months before the study,
* Treated with drugs acting on visceral fat mass &inflammation : corticosteroids, neuroleptics, alpha et beta blockers, anti-HIV tritherapy, anti-TNF alpha, antidepressant or anticoagulating agents,
* Treated with antibiotics in the 3 months prior to selection,
* With significant change in food habits or in physical activity in the 6 months before the V0 visit,
* With significant changes in lipid abnormality of antihypertensive treatment within 3 months prior to selection,
* With a personal history of bulimia or significant eating disorders according to the investigator,
* Consuming more than 3 standard drinks of alcoholic beverage daily for men or 2 daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study,
* Consuming tobacco more than 10 mg of nicotine per day
* Consuming drugs,
* Patients who suffer from claustrophobia,
* Patients who have contraindications to perform an MRI such as pacemakers, intracranial clips incompatible with MRI, heart valves, hearing aid,... and other types of implants incompatible with MRI,
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Impossible to contact in case of emergency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Absolute change of visceral fat mass (in cubic millimeter) assessed by Magnetic Resonance Imaging | between week 0, week 9, week 12

SECONDARY OUTCOMES:
Change of visceral fat mass in percentage assessed by Magnetic Resonance Imaging | between Week 0, Week 9 and Week 12
Changes of total abdominal fat mass in cubic millimeter assessed by Magnetic Resonance Imaging | between Week 0, Week 9 and Week 12
Changes of subcutaneous fat mass in cubic millimeter assessed by Magnetic Resonance Imaging | between Week 0, Week 9 and Week 12
Changes of total abdominal fat mass in percentage assessed by Magnetic Resonance Imaging | between Week 0, Week 9 and Week 12
Changes of subcutaneous fat mass in percentage assessed by Magnetic Resonance Imaging | between Week 0, Week 9 and Week 12
Changes of body fat mass measured by Dual-energy X-ray absorptiometry | between Week 0 and Week 12
Changes of body lean mass measured by Dual-energy X-ray absorptiometry | between Week 0 and Week 12
Changes of trunk fat assessed by Dual-energy X-ray absorptiometry | between Week 0 and Week 12
  calculated trunk fat
Changes of anthropometrics measurements : weight | between Week 0 and Week 12
  Weight
Changes of anthropometrics measurements : BMI | between Week 0 and Week 12
  BMI
Changes of anthropometrics measurements: Waist circumference | between Week 0 and Week 12
  Waist Circumference
Changes of anthropometrics measurements: Hip Circumference | between Week 0 and Week 12
  Hip Circumference
Changes of anthropometrics measurements: Waist to Hip ratio | between Week 0 and Week 12
  Waist to Hip ratio
Changes of anthropometrics measurements: Waist to Height ratio | between Week 0 and Week 12
  Waist to Height ratio

CONTACTS AND LOCATIONS:
Overall Officials: Marie Déciron, MD, Principal Investigator — BioFortis
Locations (6):
- France (5):
  - CEN Experimental, Dijon
  - Eurofins Optimed, Gières
  - Institut Pasteur de Lille, Lille
  - CIC Pitié Salpêtrière, Paris
  - Biofortis, Saint-Herblain
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No